CLINICAL TRIAL: NCT02565849
Title: Early Detection of Changes in Ventilatory Mechanics in Patients With Sickle Cell Anemia
Brief Title: Study of Ventilatory Mechanics in Patients With Sickle Cell Anemia
Acronym: SCA
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Cirlene Marinho, Study of Ventilatory Mechanics in Patients With Sickle Cell Anemia, Rio de Janeiro State University
Other Study IDs: EAF-8421
Record Dates: First submitted 2015-08-22; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control group: Recruited volunteers aged above 18 years with no history of smoking or hospitalization in the last three months without cardiac dysfunction, orthopedic or lung.
- Sickle Cell Anemia normal spirometry: Recruited patients aged above 18 years with no history of smoking or hospitalization in the last three months, ability to independent ambulation and spirometry tests and plethysmography with normal medical report.
- Sickle Cell Anemia spirometry abnormal: Recruited patients aged above 18 years with no history of smoking or hospitalization in the last three months, ability to independent ambulation and spirometry tests and plethysmography with altered medical report.

SUMMARY:
The Sickle Cell Anemia (SCA) is a recessive genetic condition, monogenic, resulting in defects in the red cell structure. In the investigators' country, this disease affects about 3,000 children each year and is considered one of the most prevalent disorders among the group of existing hereditary diseases.

The lungs are frequently affected in this disease by Acute Chest Syndrome (STA). Besides being the leading cause of death and the second leading cause of hospitalization in SCA, the STA is correlated with cognitive impairment frame these patients, resulting secondary Stroke vaso-occlusion of capillaries that supply the brain tissue.

Traditional tests of pulmonary function allow assess whether the person has any commitment in the respiratory system, whether obstructive, restrictive or mixed. To run these tests it is necessary that the patient understands and performs a forced expiratory maneuver to obtain reliable results. In the particular case of SCA, performing these tests it is very difficult due to the presence of cognitive impairment of varying degrees. This results in underdiagnosis of early changes in the lung parenchyma during the therapeutic window, committing the proper monitoring and treatment offered to these patients.

DETAILED DESCRIPTION:
The aim of the present study is to observe the use of the Forced Oscillation Technique (FOT) in the detection of the alterations of the respiratory mechanical in subjects with Sickle Cell Anemia. One group of patients with Sickle Cell Anemia was compared with a volunteers group without pulmonary alterations.

The experimental phase of this research was developed from the University Hospital of the Pulmonology Department Pedro Ernesto (HUPE) and Laboratory Instrumentation Biomedical of Rio de Janeiro State University (UERJ) and was approved by the Committee for Ethics in the Hospital Survey. The Informed Consent was obtained from all volunteers and patients. The study protocol complies with the Helsinki Declaration and Resolution CNS 466/12.

Patients were recruited from the Hematology clinic of the University Hospital Pedro Ernesto. After screening of the inclusion criteria, these individuals were referred to the following tests: Respiratory Function Support and Technical by Forced Oscillations.

The Respiratory Function Test were performed in the Pulmonary Function Testing Laboratory at the University Hospital Pedro Ernesto and obeyed the standard protocol of the American Thoracic Society / European Respiratory Society (ATS / ERS).

In clinical exams with the FOT, the volunteers remained seated, his head in the neutral position and used a nose clip. They were asked to maintain a basal respiration throughout the examination period through a silicone nozzle, with cheeks sustained by the hands in order to reduce the shunt effect. The system applies sinusoidal pressure signals emitting oscillatory waves in the frequency range 4-32 Hz. The results to be considered suitable, should apre sit coherence function ≥ 0.9. Three measurements were performed for 16 seconds, with rest interval between them. Finally, to analyze the parameters measured, obtained was the average of all the results. Among the parameters evaluated the resistive and reactive parameters of the respiratory system were studied, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Typing of Hemoglobin SS

Exclusion Criteria:

* History absence of respiratory infections and hospitalized in the last three months
* Asthma , smoking, rheumatological and oncological diseases, acute pain and inability to independent ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sickle cell anemia, type of hemoglobin SS, above 18 years of age, accompanied by the Hematology Clinic at the University Pedro Ernesto hospital and no contraindications for study participation
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
spirometrics parameters of pulmonary function tests assessed by forced expiratory volume in one second (FEV1) | 1 day
spirometrics parameters of pulmonary function tests assessed by forced vital capacity (FVC) | 1 day
spirometrics parameters of pulmonary function tests assessed by ratio forced expiratory volume in one second and forced vital capacity (FEV1 / FVC) | 1 day
spirometrics parameters of pulmonary function tests assessed by FEF max (Flow Forced Expiratory maximum) | 1 day
plethysmographics parameters of pulmonary function tests assessed by Total Lung Capacity (TLC) | 1 day
plethysmographics parameters of pulmonary function tests assessed by functional residual capacity (FRC) | 1 day
plethysmographics parameters of pulmonary function tests assessed by residual volume (RV) | 1 day
plethysmographics parameters of pulmonary function tests assessed by Ratio Residual Volume and Total Lung Capacity (RV / TLC) | 1 day
plethysmographics parameters of pulmonary function tests assessed by Airway resistance (Rva) | 1 day
diffusion parameters of pulmonary function tests assessed by Diffusing Capacity Carbon monoxide (DLCO) | 1 day
diffusion parameters of pulmonary function tests assessed by VA (Volume Alveolar) | 1 day
diffusion parameters of pulmonary function tests assessed by diffusion coefficient (DLCO / VA) | 1 day
forced oscillation technique assessed by zero resistance at the intercept (R0) in cmH2O/l/s | 1 day
forced oscillation technique assessed by resistance at 4 Hz (Rrs4Hz) in cmH2O/l/s | 1 day
forced oscillation technique assessed by average resistance (Rm) in cmH2O/l/s | 1 day
reactive parameters of the forced oscillation technique assessed by mean reactance (Xm) in cmH2O/l/s is a parameter related to the inhomogeneity of the respiratory system | 1 day
reactive parameters of the forced oscillation technique of the respiratory system compliance was measured by dynamic compliance (Crs, dyn) in cmH2O | 1 day
reactive parameters of the forced oscillation technique of total mechanical loading of the respiratory system was assessed using the absolute value of the respiratory impedance (Z4Hz) in cmH2O/l/s | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Cirlene Marinho, Principal Investigator — University Hospital Pedro Ernesto